CLINICAL TRIAL: NCT05974709
Title: Factors Affecting Sleep Quality in Office Workers: A Cross-Sectional Study Investigating Pillow and Mattress Factors and Musculoskeletal Symptoms.
Brief Title: Factors Affecting Sleep Quality in Office Workers
Status: Completed | Type: Observational
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Ceyhun Türkmen, Asst. Prof, Çankırı Karatekin University
Other Study IDs: 0f0534f00fdd44cc
Record Dates: First submitted 2023-07-13; First posted 2023-08-03 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Sleep; Work Related Stress; Musculoskeletal Pain; Physical Inactivity; Demographies, Family
Keywords: Sleep quality; Office workers; Sleep environment; Physical activity; Sociodemographic factors
MeSH Terms: conditions — Occupational Stress; Musculoskeletal Pain; Sedentary Behavior; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Office Workers: The study will document the sociodemographic attributes of the participants, encompassing variables such as age, gender, height, weight, educational attainment, marital status, occupation, daily working hours, and professional experience. The data pertaining to the variables in question were obtained through employment of a structured questionnaire.

SUMMARY:
This study will focus on the relationship between pillow and mattress factors, musculoskeletal disorders and sleep quality in office workers. Sleep is vital to physical and mental health, and poor sleep can negatively affect cognitive function and workplace performance. Office workers, who often work in sedentary jobs, are particularly prone to sleep disorders. Recognizing the factors that contribute to poor sleep in this population is crucial for developing interventions to improve sleep quality.

The study used a cross-sectional design and will collect data from an appropriate sample of office workers (Approximately 600 participants). Various variables will be assessed, including sociodemographic characteristics, sleep-related factors (to be measured using the Pittsburgh Sleep Quality Index), pillow characteristics, mattress-related factors, musculoskeletal symptoms, and physical activity levels (to be measured using the International Physical Activity Questionnaire).

Descriptive statistics and multiple regression analysis will be performed to analyze the data and identify factors affecting sleep quality. Fixed fixes for potential confounders and modifiers. The study aims to identify specific components of the sleep environment related to sleep disorders.

The findings of this study will contribute to the understanding of how pillow and mattress factors, along with other variables, affect sleep quality in office workers. The results may provide information for interventions aimed at improving sleep habits, optimizing the sleep environment, and improving overall well-being in this population. As a result, promoting good sleep health among office workers can have positive effects on productivity, safety and overall quality of life.

DETAILED DESCRIPTION:
INTRODUCTION

Sleeping is an important part of human life, but there is still a lot of mystery surrounding the relationship between the brain and the process of sleeping. Recent research has concluded that sleeping has much more impact on the brain than previously thought, as it resets itself and removes toxic waste byproducts which may have accumulated throughout the day. Sleeping improves memory recall, helps regulate the metabolism in the body, and reduces mental fatigue. Chronic sleep loss is a serious concern, as it can be constrained by the lack of sleep.

Sleep plays a critical role in physical health, regulating immune system functions and reducing the risk of infections. Poor sleep can weaken immune function, making individuals more susceptible to illnesses. Over the past decade, research has shown that disturbances of sleep, including insomnia complaints and extremes of sleep duration, adversely influence the risk of infectious and inflammatory disease and contribute to all-cause mortality. These findings have substantial public health implications, as 25% of the population report insomnia complaints and 10% meet diagnostic criteria for chronic insomnia. Behavioral treatments have robust efficacy, with remission of insomnia sustained in the long term. Research on sleep and health has focused on the biological mechanisms underlying these effects, which could identify those at greatest risk for adverse health consequences or be targeted to attenuate or even prevent morbidity. Furthermore, sleep is intricately linked to physical health and vitality. It contributes to the restoration and repair of various bodily systems, including the cardiovascular, musculoskeletal, and metabolic systems. Sleep loss is a common condition in developed countries, with people sleeping on average 6.8 hours per night, 1.5 hours less than a century ago. Recent epidemiological studies have revealed relationships between sleep deprivation and hypertension, coronary heart disease, and diabetes mellitus. Sleep loss has been linked to hypertension, coronary heart disease, and diabetes mellitus.

Office workers, who typically engage in sedentary work activities and spend a significant portion of their day in indoor environments, are particularly prone to sleep disturbances. Sedentary behavior is becoming an important risk factor for poor health and mortality. Population research has found that as sitting or television viewing time increases, there is an increased cardiometabolic risk, independent of moderate/vigorous physical activity (MVPA). High accelerometer-determined sedentary time has been linked to metabolic and cardiovascular risk factors in healthy adults, and prolonged or uninterrupted sedentary time has been found to be a risk factor for poor health. With the evolution of the "technology age", sedentary time is reported to be increasing due to the shift towards reduced MVPA required in occupations traditionally requiring MVPA and the increasing percentage of office workers employed in low-activity occupations. While sedentary office workers may be less exposed to many of the hazards associated with more physically demanding occupations, they may gain less of the beneficial MVPA and be exposed to more of the potentially detrimental prolonged and uninterrupted sedentary behavior.

Office workers who have sleep issues may face significant effects on their daily functioning and general quality of life. Insufficient or poor quality sleep can affect cognitive function, including the ability to pay attention, concentrate, solve problems, and make decisions. This can lower productivity, increase errors and accidents, and decrease job performance and satisfaction. Furthermore, it can have a significant impact on mental health, including an increased risk of anxiety, depression, and emotional instability. Sleep habits and workplace behaviors have a significant impact on employee performance, safety, and health, as well as organizational-level success. It is important to understand how sleep habits and sleepiness impact workers and the organization and to emphasize the impact of good sleep on productivity and safety.

Recognizing the importance of sleep and the unique challenges that office employees encounter is critical for resolving sleep disorders in this demographic. Understanding the factors that contribute to poor sleep quality among office employees allows for the development of interventions that encourage good sleep habits, optimize the sleep environment, and improve overall well-being. Education on sleep hygiene, promotion of physical exercise and mobility breaks during the workday, ergonomic workstations, and improved lighting conditions in office environments are some of the targeted measures. Office workers can improve their cognitive functioning, physical health, and general quality of life by emphasizing sleep health. Sleep problems are linked to accidents, productivity losses, and increased healthcare utilization, resulting in $15 billion in healthcare costs each year 15. Poor quality sleep can lead to accidents, productivity losses, and increased healthcare utilization.

Sleep disturbances are widespread among office workers, and recognizing the factors that contribute to these disturbances is critical for devising effective therapies to improve sleep quality in this population. The sleep environment, including pillow and mattress features, has a major impact on sleep quality.

Pillows and mattresses are important sleep environment components that have a direct impact on sleep posture, comfort, and spinal alignment. The selection of an appropriate pillow and mattress is critical for supporting the natural curvature of the spine and ensuring optimal comfort when sleeping. Inadequate pillow and mattress qualities can cause discomfort, pain, and sleep disruptions. Mattress firmness plays a leading role in reducing pain in individuals complaining of back pain. Companies are promoting mattresses with therapeutic properties, but this is not supported by sufficient evidence.

The height of a pillow is an important aspect that influences head and neck alignment during sleeping. Increasing the pillow height dramatically raises the cranial and cervical mean and peak pressures, as well as the extension and lordosis of the cervical spine. An incorrect pillow height can cause incorrect cervical spine posture, producing tension in the neck muscles and contributing to sleep-related neck pain. Similarly, the pillow's hardness or firmness can affect the support supplied to the head and neck. A pillow that is overly soft or too firm may not give enough support, causing pain and disrupting sleep.

Another important feature of pillows and mattresses is ergonomic support. Ergonomic pillows are designed to give ideal head, neck, and spine support and alignment, reducing the risk of musculoskeletal discomfort and promoting improved sleep posture. Mattresses that possess suitable firmness and support aid in maintaining spinal alignment and distributing pressure, thereby promoting a more comfortable and restorative sleep. Studies have indicated that individuals who utilize pillows and mattresses with inadequate features are at a higher risk of encountering discomfort, pain, and disruptions in their sleep patterns. The sleep quality of office workers can be enhanced by choosing pillows and mattresses that provide adequate support and comfort. This holds particular significance owing to the considerable duration of time spent in office environments, where sedentary behaviors prevail. Comprehending the influence of the aforementioned factors and enhancing the sleep environment can facilitate the advancement of superior sleep and holistic welfare.

The present research aims to examine the relationship between various pillow and mattress factors, musculoskeletal discomfort, and sleep quality in individuals working in office environments. By conducting an examination of various variables including pillow characteristics, sleep-related factors, musculoskeletal symptoms, physical activity level, and mattress-related factors, the research can identify the particular components of the sleeping environment that are most relevant to disturbances.

METHODS Study Design and Participants The purpose of this cross-sectional study was to look at the variables influencing office workers' sleep quality. Participants were gathered using a convenience sample technique from diverse workplace environments. To establish the ideal sample size, a power analysis was performed using G*Power software. The statistical test of choice was multiple regression analysis, and the computation used an effect size of f2 = 0.15. The power analysis showed that a minimum sample size of 400 participants would be needed to detect the indicated effect size with a significance level (alpha) of 0.05 and a target power (1 - β) of 0.80.

Data Collection Self-report questionnaires and objective assessments were combined to acquire the data. An extensive questionnaire including sociodemographic details and sleep-related questions was given to participants.

Sociodemographic Characteristics The study documented the sociodemographic attributes of the participants, encompassing variables such as age, gender, height, weight, educational attainment, marital status, occupation, daily working hours, and professional experience. The data pertaining to the variables in question were obtained through employment of a structured questionnaire.

Sleep-Related Variables The dependent variable will utilize to evaluate the quality of sleep was the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a frequently employed self-administered survey that assesses diverse dimensions of sleep quality and disruptions within a duration of one month. Superior scores are indicative of inferior quality of sleep. The PSQI was administered to the participants in order to obtain a comprehensive evaluation of their sleep quality.

Pillow Characteristics The study will evaluate various pillow-related variables of the participants, such as pillow height, pillow firmness, pillow composition (e.g., feather, memory foam), and pillow ergonomics. The variables were acquired via self-report inquiries, enabling participants to furnish details regarding their individual pillow predilections.

Mattress-Related Factors. Variables for mattresses include the type of mattress, such as spring or sponge, the firmness level and the degree of comfort. Participants will provide self-reported data on the above-mentioned variables to assess their personal perceptions of mattress-related factors that could potentially affect their sleep quality.

Musculoskeletal Symptoms The Nordic Musculoskeletal Questionnaire will be used to collect data on pain experienced by individuals. Specifically, the survey documents the occurrence of pain at nine different sites over the previous 12 months. Additionally, if there is pain, a rating of 1 to 10 is given.

Physical Activity Level:

Researchers will use the International Physical Activity Questionnaire (IPAQ) to assess the physical activity levels of study participants. The International Physical Activity Questionnaire (IPAQ) is a reliable and valid tool used to assess the frequency, duration and intensity of physical activity in different areas such as work, leisure and transportation. These data will facilitate capturing the potential impact of physical activity on sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be office workers.
* Participants should be at least 18 years old.
* Participants should have a minimum employment duration or professional experience.
* Participants should be willing to provide informed consent to participate in the study.
* Participants should be able to understand and complete the self-report questionnaires accurately.

Exclusion Criteria:

* Individuals who are not office workers (e.g., manual laborers, non-office-based professionals) would be excluded.
* Individuals under the age of 18 would be excluded.
* Individuals with cognitive impairments or communication difficulties that prevent them from accurately completing the self-report questionnaires would be excluded.
* Individuals who are unable or unwilling to provide informed consent would be excluded.
* Individuals with pre-existing sleep disorders or medical conditions that significantly impact sleep quality would be excluded, as they may confound the study results.
* Pregnant women or individuals with significant health conditions that affect sleep (e.g., sleep apnea, chronic pain) excluded to minimize confounding variables.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Office workers from diverse workplace environments, aged 18 years and above, with a minimum employment duration or professional experience, who are willing to participate in the study and able to understand and complete the self-report questionnaires accurately.
Sampling Method: Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Five minutes
  The Pittsburgh Sleep Quality Index is a comprehensive tool used to assess various aspects of sleep quality. It consists of 19 items, each scored on a 0-3 interval scale. These items are designed to measure subjective sleep quality, sleep latency (time taken to fall asleep), sleep duration, habitual sleep efficiency (the percentage of time spent asleep while in bed), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  To determine the overall sleep quality, the scores of these seven components are added together, resulting in a composite score that ranges from 0 to 21. Lower scores indicate better sleep quality.
Pillow height | Two minutes
  The pillow height of the office workers was recorded in cm.

SECONDARY OUTCOMES:
Mattress type | Two minutes
  The variables pertaining to mattresses encompassed the type of mattress, such as spring or foam.
Musculoskeletal Symptoms | Five minutes
  The Nordic Musculoskeletal Questionnaire was utilized to gather data pertaining to pain experienced by individuals. Specifically, the questionnaire documented the occurrence of pain in nine distinct regions over the course of the previous 12 months. Additionally, if pain was present, a rating on a scale of 1 to 10 was assigned. High scores indicate high pain.
Physical Activity Level | Five minutes
  The researchers utilized the International Physical Activity Questionnaire (IPAQ) to assess the physical activity levels of the study participants. The International Physical Activity Questionnaire (IPAQ) is a reliable and valid tool used to evaluate the frequency, duration, and intensity of physical activity in different domains such as work, leisure, and transportation. This data facilitated the capture of the potential impact of physical activity on the quality of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Ceyhun Türkmen, PhD, Principal Investigator — Çankırı Karatekin University
Locations (1):
- Çankırı Karatekin University, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Herculano-Houzel S. Neuroscience. Sleep it out. Science. 2013 Oct 18;342(6156):316-7. doi: 10.1126/science.1245798. No abstract available. PMID 24136954
- [Result] Morin CM, LeBlanc M, Daley M, Gregoire JP, Merette C. Epidemiology of insomnia: prevalence, self-help treatments, consultations, and determinants of help-seeking behaviors. Sleep Med. 2006 Mar;7(2):123-30. doi: 10.1016/j.sleep.2005.08.008. Epub 2006 Feb 3. PMID 16459140
- [Result] DeVocht JW, Wilder DG, Bandstra ER, Spratt KF. Biomechanical evaluation of four different mattresses. Appl Ergon. 2006 May;37(3):297-304. doi: 10.1016/j.apergo.2005.07.002. Epub 2005 Sep 19. PMID 16169512
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Pilcher JJ, Morris DM. Sleep and Organizational Behavior: Implications for Workplace Productivity and Safety. Front Psychol. 2020 Jan 31;11:45. doi: 10.3389/fpsyg.2020.00045. eCollection 2020. PMID 32082218